CLINICAL TRIAL: NCT05638971
Title: Optical Detection Infiltration/Extravasation in Neonates, a Continuous Monitoring for Peripheral Venous Accesses.
Brief Title: Optical Detection Infiltration/Extravasation in Neonates (ODINE)
Acronym: ODINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, D ANDREA VITO, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 3886
Record Dates: First submitted 2022-11-16; First posted 2022-12-06 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Extravasation Injury; Infant, Premature, Diseases
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sensor Group (Experimental): The first half sample size Peripheral intravenous canula will be enrolled in a non-alarming group. ivWatch will monitor the Peripheral intravenous canula insertion site collecting data without notifications. The goals of the study on the nonalarming group are: a) to evaluate ivWatch sensitivity to detect infiltration in comparison with nurse standard of care; b) to estimate the difference in terms of time to detection of ivWatch in comparison with nurse standard of care
  Interventions: Device: ivWatch

INTERVENTIONS:
Device: ivWatch — The second half sample size PIVC will be enrolled into an alarming group. ivWatch will monitor the PIVC insertion site collecting data and sending visual and auditory notifications of any infiltration. The goals of the study on the alarming group are: a) to estimate the notification rate (the number of detected infiltration in the studied period; b) to evaluate the extension and severity of the detected infiltration at the time of the notification, so to gather if ivWatch is helpful in early diagnosis
  Other Names: Sensor Allarm Group

SUMMARY:
Peripheral intravenous (PIV) therapy is one of the most common invasive procedures performed in hospitals. PIV failures often occur when fluids leak out of the vein into surrounding tissue. This failure is usually called infiltration if the leakage involves non-vesicant solutions or extravasation in case of vesicant solutions. In this clinical study both infiltration and extravasation events are indicated by the term "infiltration".

neonatal intensive care unit patients are an high-risk population for infiltration due to their intrinsic characteristic: poor and fragile vein asset, frequent and uncontrolled movements, need for prolonged intravenous drug and fluid administration. Current nursing practice involves regular PIV site assessments for continuous infusions; particular attention is payed to the identification of swelling, pain, redness, warmth, or coolness. As infiltration represents a leading cause of iatrogenic injury, an early identification, an early identification can minimize its consequences.

The ivWatch Model 400 is a device that assists medical professionals in monitoring patients for PIV infiltrations using an optical sensor. This device received FDA clearance and European Conformity Mark for use in the adult and pediatric age groups. ivWatch enhanced the Model 400 to support a new disposable electronic sensor (SmartTouch sensor). In this study, the SmartTouch Sensor will be tested in a neonatal population in a NICU setting. The new sensor design includes optical components in the sensor package, similar to a typical pulse oximeter.

Primary study objective is to investigate whether the ivWatch SmartTouch sensor may be helpful in early identification of any kind of infiltration, if compared with our current standards of care.

ELIGIBILITY:
Inclusion Criteria:

* Term and pre-term infants;
* birth weight > 1.5 kg;
* need for continuous IV therapy with an expected duration > 24 hours.

Exclusion Criteria:

* birth weight </= 1.5 kg;
* non continuous IV therapy;
* IV therapy expected duration </= 24 hours;
* skin disorders.

Ages: 0 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-05 (Actual); Study Completion 2022-07-12 (Actual)

PRIMARY OUTCOMES:
TIME | through study completion, an average of 30 hours
  How many times the ivWatch detect infiltrations before nurses. The degree of injury is calculated on the Millian scale.

SECONDARY OUTCOMES:
TIME 2 | through study completion, an average of 30 hours
  time to detection (nurse vs ivWatch) and notification rate of the ivWatch

CONTACTS AND LOCATIONS:
Locations (1):
- FPGemelliIRCCS, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallis MC, McGrail M, Webster J, Marsh N, Gowardman J, Playford EG, Rickard CM. Risk factors for peripheral intravenous catheter failure: a multivariate analysis of data from a randomized controlled trial. Infect Control Hosp Epidemiol. 2014 Jan;35(1):63-8. doi: 10.1086/674398. Epub 2013 Dec 2. PMID 24334800
- [Background] Helm RE, Klausner JD, Klemperer JD, Flint LM, Huang E. Accepted but Unacceptable: Peripheral IV Catheter Failure. J Infus Nurs. 2019 May/Jun;42(3):151-164. doi: 10.1097/NAN.0000000000000326. PMID 30985565